CLINICAL TRIAL: NCT02516436
Title: A Randomized, Double-blind, Active Control Evaluation of the Safety of BioErodible MucoAdhesive (BEMA®) Buprenorphine NX for Buprenorphine Induction of Opioid Dependent Subjects
Brief Title: The Safety of Using Buprenorphine With Naloxone in a Buccal Film to Initiate Treatment of Opioid Dependent Subjects
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: FDA did not require a clinical trial for indication.
Sponsor: BioDelivery Sciences International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BNX-302
Record Dates: First submitted 2015-08-03; First posted 2015-08-05 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Opioid Dependence
Keywords: Bunavail; Suboxone; Heroin; Zubsolv; Buprenorphine; Naloxone; Opioids; Addiction; Induction
MeSH Terms: conditions — Opioid-Related Disorders; Behavior, Addictive | interventions — Buprenorphine, Naloxone Drug Combination; Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BEMA Buprenorphine NX (Experimental): Buprenorphine with naloxone in a buccal film
  Interventions: Drug: BEMA Buprenorphine NX
- Buprenorphine (Active Comparator): Buprenorphine in a buccal film
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: BEMA Buprenorphine NX — Buprenorphine with naloxone
  Other Names: Bunavail
  Arms: BEMA Buprenorphine NX
Drug: Buprenorphine — Buprenorphine
  Arms: Buprenorphine

SUMMARY:
A randomized, double blind, active controlled study in approximately 40 opioid dependent subjects. Study duration is up to five days and includes a maximum of 3 days confinement in the clinic. Opioid dependent subjects who provide informed consent meet all entry criteria are eligible for enrollment into the study.

DETAILED DESCRIPTION:
A randomized, double blind, active controlled study in approximately 40 opioid dependent subjects. The study includes a Screening period of up to 3 days and a 2-day, double blind induction phase (subjects confined to the clinic). Screening and the first day of treatment (Day 1) may occur on the same day or Screening may occur up to 3 days prior to Day 1.

Opioid dependent subjects who provide informed consent at the Screening visit; have a Clinical Opiate Withdrawal Scale (COWS) total score ≥12; and meet other entry criteria are eligible for enrollment into the study. Subjects will be confined to the clinic beginning on Day 1 (optional confinement on Day -1) and will remain there for up to 48 hours after administration of the first study drug dose.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent obtained prior to any study procedure being performed
2. Pre-specified plan for continued treatment following study participation
3. Male or non-pregnant and non-nursing female. A female of childbearing potential is eligible to participate in this study if she is not pregnant and is using an acceptable method of birth control.
4. Subject is aged 18 to 55 years, inclusive
5. Current diagnosis of opioid substance use disorder per the Diagnostic and Statistical Manual of Mental Disorders - 5th edition (DSM-5)
6. Clinical opioid withdrawal scale (COWS) total score ≥12 prior to dosing on Day 1
7. Subject is otherwise in good general health in the judgment of the Investigator as determined from the physical and oral examination findings.
8. Subject is committed to getting help for their opioid dependence, in the judgment of the Investigator.
9. Subject has at least 1 verified contact.

Exclusion Criteria:

1. Inability to meet study participation requirements, including a stay of up to 2 nights in the clinic
2. Positive buprenorphine or methadone result on urine drug screen at Screening or Baseline
3. Concurrent Diagnostic and Statistical Manual of Mental Disorders - 5th edition diagnosis of substance use disorder (excluding opioids and tobacco)
4. Prolonged QT interval by medical history, family history, or current electrocardiogram (ECG) finding
5. History of clinically significant hepatic impairment as determined by the Investigator.
6. Use of any medication, nutraceutical or herbal product with CYP3A4 inhibition or induction properties within the past 30 days. This exclusion also extends to grapefruit juice and grapefruit juice-containing products as well as St. John's wort and St. John's wort-containing products (prescription or nonprescription drugs, vitamins, minerals, or dietary/herbal supplements).
7. Use of an investigational drug or device within the last 30 days
8. History of hypersensitivity, allergy, or intolerance to buprenorphine or naloxone
9. Increased suicidal risk, as determined by meeting any of the following:

   * History of suicidal ideation ≤ 3 months prior to Baseline with a score of 4 (intent to act) or 5 (specific plan and intent) on the electronic Columbia Suicide Severity Rating Scale (eC-SSRS)
   * History of suicidal behavior ≤1 year prior to Baseline (actual attempt, interrupted attempt, aborted attempt and/or preparatory acts/behavior) on the electronic Columbia Suicide Severity Rating Scale (eC-SSRS)
10. Lack of motivation or a pattern of prior poor response to treatment, as judged by the investigator
11. A history or current evidence of any clinically significant disorder or any other condition which in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in COWS total score for BEMA Buprenorphine NX vs BEMA Buprenorphine NX Control | At 12 hours post inital dose
  To determine if induction of opioid dependent subjects with BEMA Buprenorphine NX results in more opioid withdrawal symptoms than induction with BEMA Buprenorphine NX Control

CONTACTS AND LOCATIONS:
Overall Officials: James G Sullivan, MD, Principal Investigator — Parkway Medical Center
Locations (3):
- United States (3):
  - Birmingham, Alabama
  - Orem, Utah
  - Salt Lake City, Utah